CLINICAL TRIAL: NCT00890383
Title: Colloids in Severe Trauma: A Multi-Center Pilot Study of "Crystalloid Only" or "Crystalloid + Colloid" Volume Resuscitation in Trauma Patients (CIST)
Brief Title: Colloids in Severe Trauma
Acronym: CIST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of the Philippines (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Dr. Rafael Consunji, Clinical Associate Professor of Surgery and Chief of Surgical ICU, Dept. of Surgery, College of Medicine, University of the Philippines, Manila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCS Sur 2007-030
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Abdominal Hypertension; Abdominal Compartment Syndrome; Severe Trauma
Keywords: trauma resuscitation; abdominal hypertension; abdominal compartment syndrome
MeSH Terms: conditions — Intra-Abdominal Hypertension; Wounds and Injuries | interventions — HES 130-0.4

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crystalloid only (No Intervention): patients will receive crystalloid fluids only for volume therapy of severe trauma
- Colloid + Crystalloid arm (Active Comparator): Goal directed volume therapy for severe trauma resuscitation
  Interventions: Drug: tetrastarch (Voluven)

INTERVENTIONS:
Drug: tetrastarch (Voluven) — Goals directed volume therapy for severe trauma resuscitation
  Other Names: Voluven
  Arms: Colloid + Crystalloid arm

SUMMARY:
Background:

Fluid resuscitation is a cornerstone of the initial management of the critically injured trauma patient yet there are numerous controversies surrounding this very common practice. As a result, these controversies have been the subject of numerous clinical trials, evidence-based guidelines and systematic reviews.

With the publication of the landmark SAFE Study the equipoise between the 2 treatments (which were representative solutions for colloid and crystalloids respectively), 4% albumin and saline, was established. This has however been brought into further doubt by the paucity of data on the use of hydroxyethylstarches (HES), which are less costly and have less side effects than albumin, in trauma. More recent findings by Gruen and colleagues have shown that as much as 5% of all trauma deaths are the result of fluid overload based on the North American fluid management model for trauma (pure crystalloid fluid management).

A meta-analysis done by Kern and Shoemaker found that supranormal fluid resuscitation with crystalloids is beneficial when given before the onset of organ failure in critically ill surgical patients. Balogh and colleagues found out that when supranormal fuid resuscitation with crystalloids was applied to victims of severe trauma, this resulted in a statistically significant increase in the incidence of mortality, multiple organ failure, intra-abdominal hypertension (IAH) and abdominal compartment syndrome (ACS). More recently, Kirkpatrick and colleagues reviewed and defined a 'secondary' ACS as a direct result of fluid resuscitation. They concluded that "excess resuscitation with crystalloid fluids might be harming patients and contributing to an increased occurrence of ACS."

This study will serve as a pilot to test the hypothesis that there will be significant differences in clinical outcomes for patients with severe trauma treated with colloid (HES) plus crystalloid and crystalloid only fluid management regimens, most notably the incidence of IAH and ACS.

It is hoped that the hybrid colloid (HES) plus crystalloid fluid management regimen will provide a means to avoid the untoward fluid overload and/or other complications of pure crystalloid fluid management and the costs/complications of albumin administration.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Body weight: more than 40 kg
* Trauma patients with onset of trauma ≤ 48h prior to assessment for inclusion in study, clinically judged to be in hemorrhagic shock by the attending surgeon and with 2 or more of the following characteristics:

  * Penetrating or blunt etiology with hemodynamic instability at ER or intra-operatively
  * Severely injured with Injury Severity Score (ISS) > 15
  * Hypotension defined as either ≥ 10mmHg change in SBP or MAP ≤ 65 mmHg or needing vasopressors (dopamine ≥ 5 mcg/kg/min or norepinephrine at any dose) at the time of admission/referral
  * Hypoperfusion defined as base deficit ≥ 4 mmol/L

Exclusion Criteria:

* Known severe congestive heart failure (EF ≤ 35%)
* Known chronic renal, liver or pancreatic disease
* Known severe respiratory diseases e.g., TB, COPD, asthma
* Known coagulopathy or bleeding tendency
* Known allergy to Hydroxyethyl starch
* Participation in a clinical drug trial within the last 2 months
* Known Pregnancy or lactation
* Severe traumatic brain injury GCS < 9
* Advanced cancer (stage IV or metastatic disease)
* Patients receiving immunosuppressive drugs
* Do-not-resuscitate status
* Advanced directives restricting implementation of the protocol
* Skeletal deformity, scarring, infection, gross contamination or previous surgery at the CVP insertion site
* Severe hypoxemia if the CVP is to be inserted in the subclavian area
* Known active gastrointestinal hemorrhage
* Concomitant drug poisoning

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Intraabdominal hypertension | 30 days

SECONDARY OUTCOMES:
abdominal compartment syndrome | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rafael J Consunji, MD MPH, Principal Investigator — University of the Philippines
Locations (2):
- Philippines (2):
  - Jose Reyes Memorial Medical Center, Manila, National Capital Region
  - East Avenue Medical Center, Quezon City, NCR